CLINICAL TRIAL: NCT04612296
Title: A Longitudinal Observational Study of Self-reported Cardiomyopathy in the Heart Hive
Brief Title: The Heart Hive - Cardiomyopathy Study
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 18IC4954
Record Dates: First submitted 2020-09-01; First posted 2020-11-02 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Cardiomyopathies; Myocarditis
MeSH Terms: conditions — Cardiomyopathies; Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Research genetic analysis — Genetic analysis of DNA extracted from saliva. Participants can opt in to receive individual results of research genetic analysis for a predefined panel of clinically actionable cardiomyopathy genes.

SUMMARY:
This is an online registry and database of patients with cardiomyopathy and myocarditis, coupled with an observational study of DCM and HCM.

DETAILED DESCRIPTION:
This study utilises The Heart Hive, an international, online registry of patients with self-reported clinically diagnosed cardiomyopathy or myocarditis, and people with a family history of cardiomyopathy, enrolled on an on-going basis. Registry participants are invited to enter self-reported demographics and health data relevant to their cardiac diagnosis into The Heart Hive online database.

Registry participants with self-reported clinically diagnosed dilated (DCM )or hypertrophic (HCM) cardiomyopathy will be recruited to an observational, prospective study entailing collection of patient-reported baseline demographic data and clinical risk factors, genotyping, and annual collection of follow up data from patients, national registries (NHS Digital) and medical records.

In the pilot phase 100 DCM and 100 HCM patients will be recruited to a validation study. Consent will be sought to access medical information from health care providers in order to compare against and confirm self-reported health information. DNA will be obtained from saliva samples and tested in-house using a panel of clinically validated known Mendelian DCM and HCM genes as a second validation of the accuracy of self-reported diagnosis and to confirm equivalent genetic architecture of DCM and HCM in direct-to-patient recruited cohorts compared to traditional centre of excellence clinic-based recruitments.

Following validation of the approach and once funding is in place for genomic studies, larger numbers of affected DCM and HCM patients will be recruited to this study from the registry of research willing participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 and over),
* Males and Females,
* Capacity to provide informed consent,
* Patients with a confirmed diagnosis of cardiomyopathy or myocarditis,
* People with a family history of cardiomyopathy confirmed in a first or second degree relative.

Note: Pregnant women are eligible. This study is observational and entirely separate from clinical care.

Exclusion criteria:

* Patients who lack capacity to consent for themselves,
* Vulnerable groups (e.g. those under 18, prisoners, those in a dependent relationship, the mentally ill).
* Patients with a confirmed history of coronary artery disease:
* who have been informed by their treating physician that their cardiomyopathy is secondary to their coronary artery disease, or
* who have undergone previous percutaneous coronary intervention or coronary bypass surgery
* History of primary valvular heart disease or congenital heart disease
* Severe, untreated or untreatable hypertension (systolic blood pressures routinely >180 mm Hg and/or diastolic blood pressures >120 mm Hg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible adult patients with dilated or hypertrophic cardiomyopathy in The Heart Hive registry
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-11-09 (Actual); Primary Completion 2024-11-09 (Estimated); Study Completion 2024-11-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with cardiovascular cause of death | 90 years
  Cardiovascular death
Number of participants with arrhythmic events | 90 years
  (ventricular fibrillation, unstable sustained ventricular tachycardia, appropriate implantable cardioverter-defibrillator delivered shock, and aborted sudden cardiac death
Number of participants with major heart failure events | 90 years
  heart transplantation, left ventricular assist device implantation, unplanned heart failure, hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: James Ware, Principal Investigator — Imperial College London; Angharad Roberts, Study Director — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Candidate variants and/or genes, de-identified sequencing data, as well as de-identified high level clinical information may be shared with other clinical laboratories and researchers through databases for the purpose of improving our understanding of the relationship between genetic changes and clinical symptoms. Examples of these types of databases are dbGAP, MatchMaker Exchange, and ClinVar.